CLINICAL TRIAL: NCT02414802
Title: Study on the Application of a Novel Aspiration Thrombectomy Device Combined With Catheter-directed Thrombolysis for the Treatment of Acute Iliofemoral Deep Venous Thrombosis
Brief Title: Study of a Novel Thrombectomy Device to Treat Acute Iliofemoral Deep Venous Thrombosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Xuzhou Medical University (Other)
Responsible Party: Principal Investigator, Qianxin Huang, postgraduate student, Xuzhou Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BL2014030
Record Dates: First submitted 2015-03-25; First posted 2015-04-13 (Estimated); Last update posted 2017-01-18 (Estimated); Status verified 2017-01

CONDITIONS: Venous Thrombosis
MeSH Terms: conditions — Venous Thrombosis | interventions — Injections; Urokinase-Type Plasminogen Activator

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Combined thrombectomy device (Experimental): A manual spiral thrombus broken suction device will be used for thrombectomy before catheter-directed thrombolysis. Ten million U of urokinase once every 4-6 hours will be used during catheter-directed thrombolysis therapy. Anticoagulation therapy will be administered via subcutaneous injection of low-molecular-weight heparin calcium (LMWH-Ca 5,000 U/12 h) at discharge
  Interventions: Device: a manual spiral thrombus broken suction device; Procedure: catheter-directed thrombolysis; Drug: low-molecular-weight heparin calcium; Drug: urokinase
- Catheter-directed thrombolysis (Other): Participants will undergo catheter-directed thrombolysis alone. A total of 100,000 units urokinase will be pulse-spray injected through the catheter once every 4-6 h. Anticoagulation therapy will be administered via subcutaneous injection of low-molecular-weight heparin calcium (LMWH-Ca 5,000 U/12 h) at discharge
  Interventions: Procedure: catheter-directed thrombolysis; Drug: low-molecular-weight heparin calcium; Drug: urokinase

INTERVENTIONS:
Device: a manual spiral thrombus broken suction device — A manual spiral thrombus broken suction device will be used for thrombectomy before catheter-directed thrombolysis
  Arms: Combined thrombectomy device
Procedure: catheter-directed thrombolysis — catheter-directed thrombolysis will be used in both arms
Drug: low-molecular-weight heparin calcium — anticoagulation therapy will be administered via subcutaneous injection of low-molecular-weight heparin calcium (LMWH-Ca 5,000 U/12 h) in both arms at discharge
  Other Names: Low-Molecular-Weight Heparin Calcium for Injection
Drug: urokinase — A total of 100,000 units urokinase once every 4-6 hours will be used during catheter-directed thrombolysis therapy
  Other Names: Urokinase for Injection

SUMMARY:
The purpose of this study is to determine whether the novel aspiration thrombectomy device combined with catheter-directed thrombolysis is effective in the treatment of acute iliofemoral deep venous thrombosis (IF-DVT).

DETAILED DESCRIPTION:
Catheter-directed thrombolysis will be performed in eligible patients with acute IF-DVT. A combined mechanical thrombectomy will be used to clear the iliac thrombi in experimental group. The immediate, mid- and long-term outcomes will be recorded. Quantitative data wiil be expressed as mean ± SD, and will be compared with independent-sample t-test or paired-sample t-test. Count data will be expressed as a ratio (or percentage), and the chi-square test or the fisher's exact test will be used for comparisons. A difference with P < 0.05 will be considered statistically significant. All statistical analyses will be performed using IBM SPSS, version 22.0 (SPSS Inc., Chicago, IL, USA).

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of iliofemoral deep venous thrombosis
* Symptoms of less than 14 days' duration
* With good function status
* A life expectancy of more than 1 year
* A low risk of bleeding

Exclusion Criteria:

* Without iliac vein thrombosis
* Anticoagulation and/or thrombolysis contraindications
* Systemic infection
* Heart, hepatic, renal function insufficiency

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2014-12; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
patency of lower extremity deep venous | up to 36 months
  participants will be followed for the duration of hospital stay and will be followed for up to 36 months by lower limb vein color Doppler ultrasonography

SECONDARY OUTCOMES:
technical success rate | intraoperation
  The ratio of successful and total number of participants
thrombus removal rate | intraoperation
  The ratio of preoperative and postoperative thrombosis amount
complications | intraoperation
  a composite outcome measure of observation of whether there is evidences of puncture site hematoma, vascular injury or vascular rupture
blood loss | intraoperation
  The volume of blood loss during operation will be recorded
improvement of clinical symptoms and signs | up to 36 months
  participants will be followed for the duration of hospital stay and will be followed for up to 36 months by clinical examinations

OTHER OUTCOMES:
incidence of postthrombotic syndrome | up to 36 months
  participants will be followed for up to 36 months to observe the incidence of postthrombotic syndrome which is associated with leg swelling, pain, ulceration

CONTACTS AND LOCATIONS:
Overall Officials: Qingqiao Zhang, PHD, Study Director — Xuzhou Medical University
Locations (1):
- Department of Interventional Radiology and Vascular Surgery, the Affiliated Hospital of Xuzhou Medical College, Xuzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No